CLINICAL TRIAL: NCT04934592
Title: Correlation Between Non-motor Symptoms and Malnutrition in Patients With Parkinson's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-376
Record Dates: First submitted 2021-05-28; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study used Mini Nutrition Assessment (MNA) , Nutrition risk screening 2002(NRS-2002) and Non-motor Symptom Quest (NMSquest) to investigate the nutritional status of patients with Parkinson's disease, to analyze the correlation between non-motor symptoms and malnutrition in patients with Parkinson's disease (PD) , and to provide evidence for clinical treatment and early nutritional intervention.

DETAILED DESCRIPTION:
Data were collected by questionnaire survey.For arkinson patients who were admitted to the facility between June 2020 and July 2021 were targeted. This study used convenience sampling and included criteria: length of stay > 24 hours; Parkinson patients who met Chinese diagnostic criteria for Parkinson's disease (2016 edition) ; willing participants and able to complete the scale. Exclusion criteria: parkinsonism caused by cerebrovascular disease, encephalitis, traumatic brain injury, complete transfusion of blood, plasma, albumin within one month, severe gastrointestinal disease, metabolic disease, and other wasting diseases; Patients with critical illness, severe cognitive impairment, and inability to communicate. The study was approved by the medical ethics committee with the informed consent of all selected individuals and their families

ELIGIBILITY:
Inclusion Criteria:

* Length of stay > 24 hours; Parkinson patients who met Chinese diagnostic criteria for Parkinson's disease (2016 edition) ; willing to participate in the study and able to complete the scale.

Exclusion Criteria:

* Parkinson's disease caused by cerebrovascular disease, Encephalitis, traumatic brain injury; patients who have received whole blood, plasma, albumin within one month; patients with severe gastrointestinal disease, metabolic disease and other wasting diseases; Patients with critical illness, severe cognitive impairment, and inability to communicate.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson in the hospital
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of nutritional risk Nutrition Assessment | Within 8 hours after admission
  Mini Nutritional Assessment (MNA) score. This scale is used to evaluate the nutritional status .MNA consists of 18 subjects, covering four aspects: anthropometric assessment, general state assessment, recent diet assessment and subjective self-assessment. The total score is 30. Malnutrition is defined as score < 17, critical state of malnutrition is defined as score 17-24, and good nutrition is defined as score > 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China